CLINICAL TRIAL: NCT07242586
Title: PS-Trauma: Udvikling af Traumebehandling Til Psykiatriske Patienter Med Psykoselidelse - et Pilotstudie.
Brief Title: PS-Trauma - Development of Trauma Treatment for Patients With Co-morbid Psychotic Disorders and Traumas
Acronym: PS-Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nikolai Albert (Other)
Responsible Party: Sponsor-Investigator, Nikolai Albert, Associate professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Organization: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-25038884
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: SCHIZOPHRENIA 1 (Disorder); Schizotypal Disorder; Post Traumatic Stress Symptoms
Keywords: First episode psychosis; Trauma; Schizophrenia; psychotherapy; prolonged exposure; EMDR
MeSH Terms: conditions — Schizotypal Personality Disorder; Wounds and Injuries; Schizophrenia | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged Exposure (Active Comparator): Prolonged Exposure (PE) Arm:
  Participants assigned to PE receive up to 12 weekly individual sessions delivered by trained clinicians following the standard PE manual. Treatment focuses on repeated, systematic confrontation with trauma-related memories (imaginal exposure) and avoided situations (in-vivo exposure) to reduce fear, distress, and maladaptive avoidance. Sessions include psychoeducation, breathing retraining, development of an exposure hierarchy, and structured review of homework assignments. Therapists monitor symptom fluctuations closely and coordinate with the OPUS clinical team. PE is provided in addition to participants' usual OPUS care, and all sessions follow predefined safety and fidelity procedures.
  Interventions: Behavioral: Prolonged Exposure
- EMDR (Active Comparator): Eye Movement Desensitization and Reprocessing (EMDR) Arm:
  Participants assigned to EMDR receive up to 12 weekly individual sessions delivered by certified EMDR therapists using the standard eight-phase protocol. Treatment targets distressing trauma memories through brief, repeated exposure combined with bilateral stimulation (e.g., eye movements or tactile taps) to facilitate adaptive information processing. Sessions include history taking, identification of target memories, assessment of negative and positive cognitions, desensitization, installation, and body scan procedures. Therapists monitor symptom changes throughout and coordinate with OPUS clinicians as needed. EMDR is provided alongside usual OPUS care, with adherence ensured through protocol-based supervision and fidelity checks.
  Interventions: Behavioral: EMDR

INTERVENTIONS:
Behavioral: Prolonged Exposure — Distinguishing Features - Prolonged Exposure (PE) Arm
  This intervention is distinguished by its exclusive reliance on systematic, therapist-guided exposure procedures grounded in emotional-processing theory. PE uses structured imaginal and in-vivo exposure to reduce avoidance and fear responses and does not employ bilateral stimulation, cognitive restructuring, or memory-processing elements characteristic of other trauma-focused approaches. The protocol follows a fixed sequence emphasizing habituation and extinction learning, making it operationally and mechanistically distinct from EMDR and from supportive or stabilization-oriented therapies used in similar clinical studies.
  Arms: Prolonged Exposure
Behavioral: EMDR — Distinguishing Features - EMDR Arm
  This intervention is distinguished by its use of the standardized eight-phase EMDR protocol, which combines brief exposure to trauma memories with bilateral sensory stimulation to facilitate adaptive information processing. EMDR does not require prolonged or repeated imaginal exposure, fear-hierarchy construction, or systematic in-vivo exposure, differentiating it from PE and other exposure-based trauma treatments. Its mechanism centers on accelerating memory reprocessing rather than habituation, and the protocol includes unique components such as cognition rating, desensitization with bilateral stimulation, installation, and body scan procedures.
  Arms: EMDR

SUMMARY:
Overview:

People with psychotic disorders frequently have a history of traumatic events such as neglect, bullying, or physical and sexual abuse. Many experience significant symptoms of post-traumatic stress, but trauma-focused treatment is rarely offered in standard psychiatric care. This pilot study investigates whether two established trauma therapies can be delivered safely and acceptably to young adults with psychotic disorders receiving care in the OPUS early-intervention program.

Objectives:

The main aim is to evaluate the feasibility and acceptability of two trauma-focused treatments-Prolonged Exposure (PE) and Eye Movement Desensitization and Reprocessing (EMDR)-in patients with psychotic disorders and post-traumatic stress symptoms. The study is not designed to test treatment efficacy but to determine whether a larger randomized controlled trial is practical.

Study Design:

This is a pilot and feasibility study. Twenty OPUS patients with a diagnosis within the schizophrenia spectrum and clinically relevant PTSD symptoms will be randomly assigned to either PE or EMDR. All participants continue their usual OPUS care while attending weekly trauma-focused therapy sessions.

Assessments:

At baseline and follow-up, participants complete clinical interviews and questionnaires assessing trauma symptoms, psychotic symptoms, functioning, well-being, recovery experiences, and possible negative effects. Instruments include the PCL-5, CAPS-5, Mini-TALE, PANSS-6, PSP, WHO-5, Brief INSPIRE-O, NEQ, and CSQ.

Primary Feasibility Outcomes:

Recruitment: At least 80% of the planned sample enrolled within 6 months.

Retention: At least 70% completing ≥12 therapy sessions.

Acceptability: Participant satisfaction measured with the Client Satisfaction Questionnaire (CSQ).

Eligibility:

Inclusion:

Age ≥18

Diagnosis within the schizophrenia spectrum (ICD-10: F20-F29)

PTSD symptom score >31 on PCL-5

Current OPUS patient

Sufficient Danish language skills

Exclusion:

Substance use that prevents participation (e.g., attending sessions intoxicated)

Severe cognitive impairment

Recent changes in antipsychotic medication (within 1 month)

Risks and Safety:

Temporary increases in PTSD symptoms may occur when beginning trauma therapy; this pattern is well documented and typically followed by improvement. Previous studies show no higher risk of serious adverse events among patients with psychosis receiving trauma treatment compared with those who do not. Participants are closely monitored, and the study team works in continuous collaboration with OPUS clinicians. If a participant experiences significant clinical deterioration, the therapy can be paused or stopped, and supportive measures will be provided.

Potential Benefits:

Participants may experience a reduction in trauma-related symptoms and gain access to a treatment that is not otherwise routinely offered to patients with psychotic disorders. The study may help improve future care for this underserved population.

Funding:

The study is funded by the Nektar Foundation and conducted at the CORE Research Unit, Mental Health Services Copenhagen.

DETAILED DESCRIPTION:
This pilot study evaluates the feasibility, acceptability, and procedural integrity of delivering trauma-focused psychotherapy to individuals with schizophrenia-spectrum disorders who exhibit clinically significant post-traumatic stress symptoms. Although traumatic experiences are common in this population, trauma-focused treatment remains underutilized in routine psychiatric services due to concerns regarding symptom destabilization, insufficient clinician training, and uncertainty about optimal therapeutic approaches. Emerging evidence indicates that established trauma-focused modalities-specifically Prolonged Exposure (PE) and Eye Movement Desensitization and Reprocessing (EMDR)-can be safely delivered in patients with psychosis when accompanied by close clinical monitoring. Nevertheless, feasibility and implementation data in early-intervention settings remain limited.

The present study is designed as a randomized, parallel-group feasibility trial conducted within the OPUS early-intervention program. The overarching aim is to determine whether a larger powered efficacy trial is practicable. The study systematically evaluates recruitment and retention rates, session attendance, intervention fidelity, acceptability, and the logistical compatibility of trauma-focused treatment with existing OPUS care structures. The pilot nature of the study means that statistical analyses are exploratory and focused on estimating parameters needed for the design of a subsequent definitive trial (e.g., variability of symptom change, pre-post correlations, and event rates).

Participants are randomized 1:1 to either PE or EMDR and receive up to 12 weekly individual sessions in addition to standard OPUS treatment. Therapists are certified in the respective modalities and receive protocol-specific supervision to ensure adherence. Treatment progression follows established manuals: PE focuses on imaginal and in-vivo exposure to trauma memories and avoided situations, whereas EMDR employs bilateral stimulation during structured processing of traumatic material. Both approaches incorporate ongoing risk monitoring, review of symptom trajectories, and coordination with OPUS clinicians.

Assessments are conducted at baseline and after treatment completion. Instruments include structured diagnostic interviews for trauma and psychosis, clinician-rated symptom scales, patient-reported outcomes (trauma symptoms, well-being, recovery experience), functioning measures, and standardized adverse-event reporting tools. Particular emphasis is placed on quantifying temporary symptom fluctuations often observed during trauma therapy, documenting any clinically significant deterioration, and evaluating whether such fluctuations differ across treatment arms.

Safety procedures include predetermined criteria for pausing or discontinuing therapy, rapid communication channels with OPUS teams, and access to supportive interventions when needed. Existing evidence suggests that trauma-focused treatment does not increase the risk of psychotic relapse or severe adverse events compared with non-exposed controls; the study therefore aims to replicate and refine these safety observations within the OPUS context.

Feasibility outcomes include: (1) proportion of eligible patients successfully recruited; (2) proportion of participants completing ≥12 sessions; (3) treatment adherence rated through fidelity checklists; (4) participant-reported acceptability and satisfaction; and (5) operational practicality, including therapist burden, integration with OPUS scheduling, and need for additional support structures. These metrics will inform the design parameters for a future multicenter randomized controlled trial.

Overall, this pilot study seeks to generate high-quality feasibility data on the integration of trauma-focused psychotherapy into early-intervention services for individuals with psychotic disorders. Findings will guide the refinement of recruitment strategies, safety procedures, intervention delivery, and outcome assessment protocols to support a subsequent adequately powered trial aimed at evaluating clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age Diagnosis within schizophrenia spectrum (ICD10 F2X) PTSD symptoms equivalent to above 31 on the PCL-5 Included in Early intervention services (OPUS) Talks and understands Danish

Exclusion Criteria:

* Substance or alcohol abuse interfering with the therapy Indication of sever cognitive impairment Changes in antipsychotic treatment within the last month

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recrutment | 6 months
  80% of planed participants will be included within 6 months
Retensionrate | 8 months
  A minimum of 70% of participants will conclude the therapy sessions

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Albert, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
If accepted the data will be deposited in the Danish National Archives
Supporting Information: Study Protocol, Analytic Code
Time Frame: Depending on the national Archives the data will deposited within a year of completion of the study (07.31.2027)
Access Criteria: Access to data is based on review by the Danish national archives and are not decided by the researchers
URL: https://en.rigsarkivet.dk/